CLINICAL TRIAL: NCT03030950
Title: Effects of Peri-neural Dexmedetomidine on the Pharmacodynamic Profile of Bupivacaine-induced Adductor Canal Block in Patients Undergoing Arthroscopic Medial Meniscectomy
Brief Title: Perineural Dexmedetomidine in Adductor Canal Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Lecturer of anesthesia and critical care medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-31-2016
Record Dates: First submitted 2017-01-19; First posted 2017-01-25 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Arthroscopic Medial Meniscectomy
MeSH Terms: interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Adductor canal block will be performed before induction of general anesthesia. Patients will be positioned in the supine position with knee slightly flexed and leg externally rotated followed by ultrasound scanning of the middle of thigh using 13-6 MHz linear array probe. The ultrasound probe will be placed over the anterior aspect of the patient's thigh, mid-point between the inguinal crease and medial femoral condyle. The scan will be focused on the femoral artery pulsations aiming to try to visualize the nerves in the adductor canal on both sides (lateral and medial) of the pulsating femoral artery. 20 ml bupivacaine 0.25% combined with 75 mcg dexmedetomidine will be injected. The study solution will be injected underneath the fascia of sartorius muscle.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Adductor canal block will be performed before induction of general anesthesia. Patients will be positioned in the supine position with knee slightly flexed and leg externally rotated followed by ultrasound scanning of the middle of thigh using 13-6 MHz linear array probe. The ultrasound probe will be placed over the anterior aspect of the patient's thigh, mid-point between the inguinal crease and medial femoral condyle. The scan will be focused on the femoral artery pulsations aiming to try to visualize the nerves in the adductor canal on both sides (lateral and medial) of the pulsating femoral artery. 20 ml bupivacaine 0.25% combined with 75 mcg dexmedetomidine will be injected. The study solution will be injected underneath the fascia of sartorius muscle.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — to investigate the effect of dexmedetomidine on motor and sensory properties of adductor canal block
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Normal saline — to give normal saline to the other group as a placebo
  Other Names: Saline
  Arms: Control group

SUMMARY:
This study is designed to explore the effects of peri-neural dexmedetomidine on the duration and motor sparing potentials of adductor canal block in adult patients undergoing arthroscopic medical meniscectomy in the setting of multimodal analgesia. The investigators ultimate goal is to increase the postoperative analgesic time and to preserve quadriceps muscle strength to promote safe and early ambulation.

DETAILED DESCRIPTION:
Peripheral nerve blocks using long-acting local anesthetics are commonly utilized as the sole anesthetic technique or as an adjuvant to general anesthesia for post-operative pain management. However, the duration of sensory block after single dose of long acting local anesthetics is not consistently sufficient to avoid the use of postoperative opioids. Many adjuvants were added to local anesthetics to augment the potency and prolong the duration of peripheral nerve blocks. Alpha-2 adrenoceptor agonists such as clonidine have been shown to increase the duration of peripheral nerve block. Dexmedetomidine is a more potent and selective α-2-adrenoceptor compared to clonidine. Peri-neural dexmedetomidine was evaluated in animal studies where it prolonged the duration of sensory and motor blocks of local anesthetics without any evidence of neurotoxicity for up to 14 days after initial administration. The effectiveness of perineural dexmedetomidine in augmenting the duration of sensory block of upper limb extremity blocks is based on good quality clinical evidence.

Arthroscopic knee surgery is associated with severe postoperative pain which could be adequately managed by femoral nerve block. However femoral nerve block has been associated with significant motor block and decreased quadriceps muscle strength which may delay ambulation and increase the risk of falling. More recently, adductor canal block (ACB) emerged as a selective motor sparing effective variant of femoral nerve block. Compared with baseline values, the adductor canal block reduces quadriceps muscle strength by 8%, versus 49% for the femoral nerve block. A recent dose finding MRI study reported that 20 ml of local anesthetic is the closest volume to the ED95 for adductor canal block with minimal proximal spread and an estimated success probability of 95.1% (95% credibility interval: 91-98%).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of aged (18-45), ASA physical status I or II undergoing arthroscopic medial meniscectomy.

Exclusion Criteria:

* Body mass index greater than 35 kg/m2.
* Pregnancy.
* Unstable coronary artery disease, congestive heart failure, or arrhythmias.
* Baseline heart rate (HR) less than 60 beats/min or baseline systolic blood pressure less than 100 mmHg.
* Pre-existing neurological deficits or neuropathy.
* Significant psychiatric or cognitive conditions interfering with consent or assessment.
* Significant renal or hepatic impairment;
* Severe bronchopulmonary disease, including chronic obstructive pulmonary disease and obstructive sleep apnea.
* Known contraindications to peripheral nerve block, including local skin infections, bleeding diathesis, and coagulopathy.
* Allergies to local anesthetics, dexmedetomidine, or any component of multimodal analgesia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours
  the time passed till the patient first analgesic request

SECONDARY OUTCOMES:
richmond agitation sedation scale | 24 hours
  A scale to assess the patient sedation and agitation
duration of sensory block | 24 hours
  The time needed to regain the patient sensation
onset of sensory block | minutes
  A blinded investigator will assess sensory block with pinprick test every 5 min for 30 min after injection of the study medication using a 3-point scale: 0 ═ complete loss of sensation, 1 ═ partial loss of sensation and 2 ═ normal sensation. Assessment will be done in comparison to contra-lateral area
blood pressure | 24 hours
  mmHg
heart rate | 24 hours
  beat per minutes
onset of motor block (by assessment of quadriceps muscle strength) | minutes
  The maximum voluntary isometric contraction (MVIC) of the quadriceps femoris muscle will be measured using a handheld dynamometer
resting visual analogue score | 24 hours
  the grade of pain during rest as experienced by the patient, rated from 0 to 10
dynamic visual analogue score | 24 hours
  the grade of pain with movement as experienced by the patient, rated from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdulatif, Professor, Study Director — Professor and member of research committee of anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No